CLINICAL TRIAL: NCT06943716
Title: A Retrospective Cohort Study Evaluating the Efficacy of Bilateral Modified Catheter Antegrade Cerebral Perfusion (Modified bACP) in Acute Type A Aortic Dissection Surgery
Brief Title: Efficacy of Bilateral Modified Catheter Antegrade Cerebral Perfusion in Acute Type A Aortic Dissection Surgery
Status: Terminated | Type: Observational
Why Stopped: Terminated due to insufficient enrollment to achieve desired statistical power. A new IRB approval will be sought to extend the retrospective data collection period.
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMUH113-REC1-183; CMUH113-REC1-183 (Other: Institutional Review Board, China Medical University Hospital)
Record Dates: First submitted 2025-04-16; First posted 2025-04-24 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Acute Type A Aortic Dissection
Keywords: Bilateral Catheter Antegrade Cerebral Perfusion; Acute Type A Aortic Dissection; Neurological Complications; Modified bACP; Retrospective Cohort

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Modified bACP Group: Patients who underwent acute Type A aortic dissection repair using the Bilateral Modified Catheter Antegrade Cerebral Perfusion (Modified bACP) technique. This observational group received the modified perfusion strategy aimed at reducing surgical trauma and enhancing cerebral protection.
  Interventions: Procedure: Modified Catheter Antegrade Cerebral Perfusion (Modified bACP)
- Conventional Perfusion Group: Patients who underwent acute Type A aortic dissection repair using the conventional brain perfusion technique (e.g., standard bilateral antegrade cerebral perfusion). This group serves as the comparison cohort for evaluating the effects of the modified technique.
  Interventions: Procedure: Conventional Brain Perfusion

INTERVENTIONS:
Procedure: Modified Catheter Antegrade Cerebral Perfusion (Modified bACP) — A modified bilateral catheter antegrade cerebral perfusion technique used for acute Type A aortic dissection repair. This approach aims to reduce surgical trauma by avoiding additional right axillary access while maintaining stable cerebral perfusion.
  Groups: Modified bACP Group
Procedure: Conventional Brain Perfusion — Patients receiving the conventional perfusion strategy for aortic arch surgery, which may include standard bilateral ACP based on the surgeon's preference and the patient's condition.
  Groups: Conventional Perfusion Group

SUMMARY:
This retrospective cohort study aims to evaluate the efficacy of a Bilateral Modified Catheter Antegrade Cerebral Perfusion (Modified bACP) technique in acute Type A aortic dissection surgery. Medical records from January 1, 2021, through October 31, 2024, at China Medical University Hospital will be reviewed. The primary outcomes include in-hospital mortality and stroke rate, while secondary outcomes include ICU/hospital stay, mechanical ventilation duration, and other postoperative complications (e.g., acute kidney injury, sepsis, myocardial infarction).

DETAILED DESCRIPTION:
Background and Rationale Acute Type A aortic dissection (ATAAD) is a life-threatening condition requiring urgent surgical repair. Prolonged circulatory arrest increases the risk of neurological complications. Bilateral antegrade cerebral perfusion (bACP) has shown potential to reduce ischemic injury. However, conventional bACP requires additional surgical access. This study examines a Modified bACP approach that may reduce surgical trauma while maintaining adequate cerebral perfusion.

Objectives This retrospective cohort study evaluates whether Modified bACP improves postoperative outcomes compared to conventional perfusion strategies in ATAAD surgery at China Medical University Hospital (2021/1/1-2024/10/31).

Methods We will collect and analyze medical records of adult patients who underwent ATAAD repair, comparing those who received Modified bACP to those managed with conventional perfusion.

Outcome Measures

Primary Outcomes:

In-hospital mortality 30-day mortality

Secondary Outcomes:

Hospital length of stay (day) ICU length of stay (day) Mechanical ventilation duration (hours) Need for tracheostomy Stroke Postoperative neurological deficit Paraplegia Coma Atrial fibrillation (Af) Myocardial infarction Acute kidney injury (AKI) Dialysis requirement Reoperation for bleeding Sepsis Significance This study aims to provide comprehensive data on the safety and efficacy of Modified bACP in ATAAD surgery, potentially improving neurological protection and reducing other major complications and resource utilization. The findings may guide clinical practice and inform future protocol developments.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ 18 years old) who underwent acute Type A aortic dissection repair at China Medical University Hospital between January 1, 2021, and October 31, 2024.

Exclusion Criteria:

* Preexisting severe neurological impairment (e.g., stroke or other major neurological deficits before surgery).
* Age < 18 years.
* Pregnant patients.
* Insufficient or missing medical records preventing data analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with acute Type A aortic dissection who underwent surgical repair at China Medical University Hospital. The population includes individuals receiving either Modified bACP or conventional perfusion during the specified period.
Sampling Method: Non-Probability Sample
Enrollment: 273 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2025-04-11 (Actual)

PRIMARY OUTCOMES:
Stroke | Through hospital discharge (on average about 14 days post-surgery)
  New-onset cerebrovascular accident or imaging-confirmed stroke during hospitalization.

SECONDARY OUTCOMES:
Postoperative Neurological Deficit | Through hospital discharge (on average about 14 days post-surgery)
  Any persistent neurological deficit (e.g., motor/sensory deficits) identified after surgery.
30-day Mortality | Assessed at 30 days post-surgery
  All-cause mortality occurring within 30 days after the surgical procedure.
Hospital Stay (day) | From end of surgery to hospital discharge (up to 21 days).
  Total number of days from the operation date to the date of hospital discharge.
ICU Stay (day) | From end of surgery to ICU discharge (up to 10 days).
  Length of stay in the intensive care unit after surgery.
Mechanical Ventilation (hour) | From end of surgery until extubation (up to 72 hours).
  Duration of mechanical ventilation in hours.
Acute Kidney Injury (AKI) | During the index hospitalization (on average about 10-14 days post-surgery)
  Acute kidney injury defined by changes in serum creatinine or urine output (e.g., KDIGO criteria).
Dialysis Requirement | During the index hospitalization (on average about 10-14 days post-surgery)
  Proportion of patients requiring renal replacement therapy (dialysis) postoperatively.
Reoperation for Bleeding | During the index hospitalization (on average about 72 hours post-surgery)
  Number of patients requiring a return to the operating room for bleeding control or hematoma.
Sepsis | During the index hospitalization (on average within 7 days post-surgery)
  Incidence of sepsis as defined by current guidelines (e.g., Sepsis-3), typically requiring positive cultures and organ dysfunction.
Atrial Fibrillation (Af) | During the index hospitalization (on average within 7 days post-surgery)
  New-onset atrial fibrillation or documented arrhythmia episodes requiring clinical management.
Myocardial Infarction | During the index hospitalization (on average about 10-14 days post-surgery)
  Clinically confirmed myocardial infarction based on ECG changes, cardiac enzymes, and clinical symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: En-Bo Wu, M.D., Principal Investigator — Department of Anesthesiology, China Medical University Hospital, China Medical University, Taichung City 404, Taiwan
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to institutional privacy policies and IRB regulations that restrict the release of patient-level data. The de-identified data are only approved for internal use by the research team and cannot be disclosed to external parties without additional ethics approval.

REFERENCES:
- [Result] Pitts L, Kofler M, Montagner M, Heck R, Iske J, Buz S, Kurz SD, Starck C, Falk V, Kempfert J. Cerebral Protection Strategies and Stroke in Surgery for Acute Type A Aortic Dissection. J Clin Med. 2023 Mar 15;12(6):2271. doi: 10.3390/jcm12062271. PMID 36983272